CLINICAL TRIAL: NCT02864004
Title: Apomorphine Pump in Early Stage of Parkinson's Disease
Brief Title: Apomorphine Pump in Early Stage of Parkinson's Disease (EARLY-PUMP)
Acronym: EARLY-PUMP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35RC15_9724_EARLY-PUMP
Record Dates: First submitted 2016-07-15; First posted 2016-08-11 (Estimated); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson disease; Quality of Life; Apomorphine infusion
MeSH Terms: conditions — Parkinson Disease | interventions — Apomorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APO group (Experimental): An apomorphine pump will be installed and adjusted. The target dose corresponds to the patient's individual optimized dose :maximum dose of 10 mg/hour for 16 hours
  Interventions: Drug: Apomorphine
- Control group (Active Comparator): Patients will be optimally treated with oral dopaminergic therapy to obtain the best medical treatment (BMT) defined as the most efficient single treatment options or their combination.
  Interventions: Other: Best Medical Treatment

INTERVENTIONS:
Drug: Apomorphine — Apomorphine (5 mg/ml) is supplied as solution for infusion in a 10 ml glass ampoule Hourly flow rate is adjusted during the whole duration of the study to doses of minimum 3 mg/hour up to a maximum of 10 mg/hour
  Other Names: Apokinon
  Arms: APO group
Other: Best Medical Treatment — Most efficient single treatment of Parkinson's disease symptoms or their combinations, in concordance with the guidelines of the European Federation of Neurological Societies
  Arms: Control group

SUMMARY:
The aim of the study is to assess the use of the apomorphine pump in earlier stages of Parkinson' Disease (PD), when motor complications have just developed and before patients are significantly affected in their social and occupational functioning. The investigators hypothesize that apomorphine pump is superior in terms of positive impact on quality of life (QoL) to oral medical therapy alone at a relatively early stage of PD, before the appearance of severe disabling motor complications thus favoring the maintain of patients' social and occupational status with a significant positive economic impact of the health system.

DETAILED DESCRIPTION:
The recruitment period will be 36 months. The duration of the study period will be one year for each patient due to:

* adjustments of apomorphine pump parameters and oral medication (3 months interval),
* motor and psychosocial changes which need time to develop and have an impact on QoL.

At the end of the study period, two additional visits at Months 18 and 24 will be performed during an long term follow up to collect QoL and costs related data required to medico-economic analysis.

APOMORPHINE (APO) group:

The apomorphine pump will be installed and adjusted at baseline during a first hospitalization (10 days). Modifications of the hourly flow of the pump and readjustment (reduction) of anti-parkinsonian oral medication will be checked and performed at Months 1, 2, 4, 5, 6, 9 during visits and phone calls, and at month 3 during a 3 days hospitalization. Clinical evaluations will be performed at months 6 and 12.

Control group:

Patients will be treated by optimized medical treatment according to the guidelines of the European Federation of Neurological Societies. Dose adjustments will be done at Months 3, 6, 9. Clinical evaluations will be performed at months 6 and 12.

In both groups, data for medico-economic evaluation will be collected from patients at baseline, Months 6, 12, 18 and 24 for Quality Adjusted Life Year (QALYs) and costs related data from a patient's diary and French Health Insurance database.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≤ 65 years,
* Idiopathic PD (According to British Brain Bank Criteria) without any other known or suspected cause of Parkinsonism,
* Hoehn and Yahr stage ≤ 2.5 in the best ON,
* Disease duration ≥ 4 years,
* Presence of fluctuations and/or dyskinesias for no more than 3 years,
* One of the two following forms of impairment :

  * Impairment in activities of daily living (MDS-UPDRS II>6) due to PD-symptoms despite medical treatment in the worst condition or,
  * Impairment of social and occupational functioning (measured with SOFAS) due to PD-symptoms despite medical treatment (51-80%),
* PDQ39 completed,
* Able to understand and remember the component of the study,
* Written informed consent,
* Patients covered with social insurance.

Exclusion Criteria:

* Dementia (MoCA < 22),
* Major uncontrolled depression at the time of assessment (BDI > 25) or Bipolar disease,
* Active hallucinations or history of hallucinations in the past year,
* Need for nursing care,
* Previous use of apomorphine pump treatment,
* History of respiratory depression,
* History of deep brain stimulation or lesional surgery for PD or intrajejunal L-Dopa,
* Presence of severe freezing or clinically relevant postural instability leading to falls during the ON state,
* Symptomatic clinically relevant and medically uncontrolled orthostatic hypotension,
* Clinically relevant hepatic dysfunction (total bilirubin >2.0 mg/dL, Alanine Amino Transferase (ALT) and Aspartate Amino Transferase (AST) >2 times the upper limit of normal),
* Clinically relevant renal dysfunction (serum creatinine >2.0 mg/dL),
* Pregnant and breastfeeding women,
* Hypersensitivity to apomorphine or any excipients of the medicinal product,
* Concomitant therapy or within 28 days prior to baseline with : alpha-methyl dopa, metoclopramide, reserpine, neuroleptics (except Clozapine), methylphenidate, or amphetamine, intrajejunal Ldopa,
* History or current drug or alcohol abuse or dependencies,
* Patients with a borderline QT interval corrected for heart rate according to Bazett's formula (QTc) of >470 ms for male and >480 ms for female at screening or history of long QT syndrome;
* Adults legally protected (under judicial protection, guardianship or supervision), persons deprived of their liberty.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Difference in the Parkinson's Disease Quality of Life Questionnaire (PDQ39) summary index between the baseline assessment and the assessment at 12 months' follow up | 12 months

SECONDARY OUTCOMES:
Change in the Patient Global Impression of Change (PGIC) | 12 months
Change in the Neurologist Global Impression of change (CGI-I) | 12 months
Change in non-motor aspects of experiences of daily living (MDS-UPDRS I) between the baseline assessment and the assessment at 12 months' follow up | 12 months
Change in motor aspects of experiences of daily in "on" and "off" medication (MDS-UPDRS II) between the baseline assessment and the assessment at 12 months' follow up | 12 months
Change in motor examination during "on" periods (MDS-UPDRS III) between the baseline assessment and the assessment at 12 months' follow up | 12 months
Change in motor complications with MDS-UPDRS IV between the baseline assessment and the assessment at 12 months' follow up | 12 months
Change in number of hours per day in the "best ON" state between the baseline assessment and the assessment at 12 months' follow up | 12 months
Change in number of hours per day in "ON" with dyskinesia between the baseline assessment and the assessment at 12 months' follow up | 12 months
Change in number of hours per day in "OFF" state between the baseline assessment and the assessment at 12 months' follow up | 12 months
Change in number of Sleeping-hours per day between the baseline assessment and the assessment at 12 months' follow up | 12 months
Change in Score of the Non-Motor Symptoms Scales (NMSS) for PD between the baseline assessment and the assessment at 12 months' follow up | 12 months
Change in psychosocial functioning PD (SCOPA-PS) between the baseline assessment and the assessment at 12 months' follow up | 12 months
Changes in score of depressive symptoms (BDI) between the baseline assessment and the assessment at 12 months' follow up | 12 months
Change in occurrence of anxiety (STAI-S) between the baseline assessment and the assessment at 12 months' follow up | 12 months
Change in pain assessed on the Visual Analog Scale (VAS) between the baseline assessment and the assessment at 12 months' follow up | 12 months
Change in cognitive function between the baseline assessment and the assessment at 12 months' follow up | 12 months
  Change in cognitive function assessed by the Neuroscience Parkinson network's (NS-PARK) battery test
Change in apathy assessed on the Apathy Scale between the baseline assessment and the assessment at 12 months' follow up | 12 months
Change in apathy assessed on the short version of Lille Apathy Rating Scale (LARS) between the baseline assessment and the assessment at 12 months' follow up | 12 months
Change of dose for treatments assessed by levodopa (L-DOPA) equivalents between the baseline assessment and the assessment at 12 months' follow up | 12 months
Change in behavioral symptoms assessed by Ardouin Scale between the baseline assessment and the assessment at 12 months' follow up | 12 months
Frequency, type and severity of therapy-related adverse events | 12 months
Skin changes assessed by a clinical exam | 12 months
Full blood count | 12 months
Epworth Sleepiness Scale | 12 months
Incremental Cost-Effectiveness Ratio (ICER) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sophie DRAPIER, Dr, Principal Investigator — Rennes University Hospital
Locations (20):
- France (20):
  - Amiens University Hospital, Amiens
  - Bayonne Côte Basque Hospital, Bayonne
  - Pellegrin University Hospital, Bordeaux
  - Pierre Wertheimer Hospital, Bron
  - Caen University Hospital, Caen
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - Lille University Hospital, Lille
  - APHM, hospital of Timone, Marseille
  - Clinique Beau-Soleil, Montpellier
  - Montpellier University Hospital, Montpellier
  - Nancy University Hospital, Nancy
  - Laennec Hospital, Nantes
  - Pasteur 2 University Hospital, Nice
  - Caremeau University Hospital, Nîmes
  - Pitié-Salpêtriere Hospital, Paris
  - Poitiers University Hospital, Poitiers
  - Rennes University Hospital, Rennes
  - Saint-Etienne University Hospital, Saint-Etienne
  - Hautepierre University Hospital, Strasbourg
  - Purpan University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No